CLINICAL TRIAL: NCT04477915
Title: The Effects of Auxiliary Respiratory Muscles Exercises and Core Stabilization Exercises on Maximum Oxygen Uptake and Pulmonary Function
Brief Title: Effects of Two Different Exercise Practices on Maximum Oxygen Uptake and Pulmonary Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KaratayUH
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Core stabilization; Auxiliary Respiratory Muscles; Maximum oxygen uptake; Pulmonary function

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core stabilization Exercise (Experimental): Core stabilization exercise include, plank, lateral plank, swimmer, flutter kick and bridge exercises. Exercises will be carried out under the supervision of a physiotherapist 3 days in a week separate time periods. Our study will take 6 weeks.
  Interventions: Other: Core exercises
- Auxiliary respiratory exercises (Experimental): Auxiliary respiratory exercises include, strengthening and stretching exercises for trapezius, sternocleidomastoideus, pectoralis major and serratus anterior muscles. exercises will be carried out under the supervision of a physiotherapist 3 days in a week separate time periods. Our study will take 6 weeks.
  Interventions: Other: Auxiliary respiratory exercises
- Control (No Intervention): Control Group

INTERVENTIONS:
Other: Core exercises — Core stabilization exercise include, plank, lateral plank, swimmer, flutter kick and bridge exercises.
  Arms: Core stabilization Exercise
Other: Auxiliary respiratory exercises — Auxiliary respiratory exercises include, strengthening and stretching exercises for trapezius, sternocleidomastoideus, pectoralis major and serratus anterior muscles.
  Arms: Auxiliary respiratory exercises

SUMMARY:
Cardiopulmonary capacities of individuals are an indication of both the individual's exercise capacity and endurance. The most important indicator of cardiopulmonary capacity is maximum oxygen uptake and respiratory parameters. Auxiliary respiratory muscles exercises and core stabilization exercises have a place in increasing the maximum oxygen uptake. There are studies investigating the effects of respiratory muscle training and core stabilization training on maximum oxygen uptake in the literature. However, there is no study in the literature comparing the effects of auxiliary respiratory muscles exercises and core stabilization exercises on maximum oxygen uptake and respiratory parameters. Thanks to the findings to be obtained from our study, it is aimed to contribute to the literature with objective, evidence-based results in this field.

DETAILED DESCRIPTION:
The study will be carried out on volunteers after the approval of the ethics committee. Before the research, individuals and / or their relatives will be informed about the purpose and content of the study. Volunteer individuals between the ages of 18-25 without any known health problems will be included in the study after obtaining their informed consent.

Participants will be randomly divided into three groups: control group, core stabilization exercises and auxiliary respiratory muscles exercises.

In the core stabilization exercises and auxiliary respiratory muscles exercises groups, exercises will be carried out under the supervision of a physiotherapist 3 days in a week separate time periods. Core stabilization exercise include, plank, lateral plank, swimmer, flutter kick and bridge exercises. Auxiliary respiratory exercises include, strengthening and stretching exercises for trapezius, sternocleidomastoideus, pectoralis major and serratus anterior muscles. Our study will take 6 weeks. The demographic information of the participants will be recorded and the VO2max values of the participants before and after the study will be measured with the H / P Cosmos Mercury Med device using the balke protocol. Respiratory function tests of participants will be measured with Cosmed Fitmate Med device before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals without any known health problems

Exclusion Criteria:

* Acute myocardial infarction, Unstable angina, Uncontrolled cardiac arrhythmias, Endocarditis, Various symptomatic aortic stenosis, Acute pulmonary embolism, pulmonary infarction and deep vein thrombosis, Acute myocarditis, pericarditis, physically not enough fit to test safely

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Maximum oxygen uptake at 6 weeks | Baseline and week 6
  the VO2max values of the participants before and after the study will be measured with the H / P Cosmos Mercury Med device using the Balke Ware protocol.
Change from baseline in Pulmonary function tests at 6 weeks | Baseline and week 6
  Forced expiratory volume in 1 second / forced vital capacity (FEV1/FVC), vital capacity and maximum voluntary ventilation (MVV) values of the participants will be measured with Cosmed Fitmate Med device before and after the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Gerçek, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)